CLINICAL TRIAL: NCT06227663
Title: Impact Assessment on Anxiety of Using a KOALOU® Digital Application for Children Undergoing Scheduled Ambulatory Surgery Compared to Those Who do Not Use the Application .
Brief Title: Impact on Anxiety of a Digital Application for Children Undergoing Scheduled Ambulatory Surgery
Acronym: KOALOU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier de Valenciennes (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021-03
Record Dates: First submitted 2022-08-29; First posted 2024-01-29 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2023-11

CONDITIONS: Anxiety Postoperative
Keywords: Preoperative anxiety; Ambulatory surgery; Pediatrics anesthesia; Digital application; Postoperative maladaptative behavioral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Access to the KOALOU(®) digital application (Experimental)
  Interventions: Behavioral: KOALOU(®) digital application
- No access (No Intervention)

INTERVENTIONS:
Behavioral: KOALOU(®) digital application — Digital app that prepares children for the ambulatory surgery care pathway by assessing their anxiety and educating them about anesthesia and surgery
  Arms: Access to the KOALOU(®) digital application

SUMMARY:
The prospect of pediatric surgery is a source of preoperative anxiety for children and their parents. It affects 50% of children waiting for surgery and the causes vary according to age. It has been shown that pre-operative anxiety in children often leads to behavioral changes. Pre-operative anxiety is often managed by pharmacological premedication. However, there are many alternative techniques to reduce children's anxiety before surgery.

The use of an application dedicated to pediatric anesthesia used from the moment of the anesthesia consultation would allow to reduce this anxiety by allowing a varied course of information involving the child in his preparation before the surgery.

First, it allows an evaluation of the pre-operative anxiety level of children via validated scales. Secondly, it provides information to the children using methods adapted to their age and level of understanding.

Thus, if this method were validated, other hospitals could use this application to develop a tool that would benefit the many children who undergo surgery each year.

ELIGIBILITY:
Inclusion criteria :

* Patients from 3 to 12 years old.
* Outpatient hospitalization for a scheduled surgery or procedure under general anesthesia.
* Clinically stable condition.
* Information note sent to parents and collection of their consent to their child's participation in the study.
* Parental affiliation to a social security system.

Exclusion criteria :

* Urgent intervention situation.
* Patient included in another study.
* No compatible hardware for the application or no internet connection (smartphone, tablet, computer).
* Patient not affiliated to social security.
* Mental retardation or psychoactive disorders.
* Intravenous induction.
* Need for premedication.
* Patient who had general anesthesia less than one year ago and/or after the age of 3.
* Patient who had surgery less than one year ago and/or after the age of 3.
* Child's refusal.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 98 (Actual)
Dates: Start 2021-08-19 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-09-22 (Actual)

PRIMARY OUTCOMES:
Preoperative anxiety in the operating room before the induction | in the operating room before the induction
  Compare the anxiety of children in the operating room before induction according to the use or not of the KOALOU® application. The primary endpoint is defined by the mYPAS-SF score calculated in the operating room before induction. The mYPAS-SF is the Yale Preoperative Anxiety Scale in his short form. It is going from 4 to 18. 4 is the minimal level of anxiety and 18 is the maximal level of anxiety.

SECONDARY OUTCOMES:
Postoperative maladaptative behavioral | during the day-7 phone call
  Compare the existence of postoperative maladaptative behavioral of children on day-7 depending on the use or not of the KOALOU® application using the PHBQ score. The PHBQ score is the Post Hospitalization Behavioral Questionnaire. It is going from 23 to 115. 23 means no postoperative maladaptative behaviors and 115 means maximum postoperative maladaptative behaviors.
Preoperative anxiety in the surgery department before the surgery | in the surgery department before the surgery
  Compare the anxiety of children in the surgery department before the surgery according to the use or not of the KOALOU® application using the mYPAS-SF score. The mYPAS-SF is the Yale Preoperative Anxiety Scale in his short form. It is going from 4 to 18. 4 is the minimal level of anxiety and 18 is the maximal level of anxiety.
Anxiety of the parents | In our hospital the chid is going alone in the operating room. The anxiety of the parents is measured in the hospitalization room after the separation with the child when the child is going in the operative room
  Compare the anxiety of the parents according to the use or not of the KOALOU® application after the separation with the child using the STAI-YA scale. The STAI-YA scale is the State Trait Anxiety Inventory in the A form. It is going from 20 to 80. 20 is the minimal level of anxiety and 80 is the maximal level of anxiety.
Acceptance of the mask | At the time of the induction
  Compare the proportion of the acceptance of the mask at the time of the induction according to the use or not of the KOALOU® application
Agitation of the child | in the postoperative monitoring room after the operation when the child is waking up. It is measured just after the entry and just before the exit of the postoperative monitoring room
  Compare the level of agitation of the child in the postoprative monitoring room according to the use or not of the KOALOU® application using the Watcha Scale score. It is going from 1 to 4. 1 means that the child and 4 that the child is agitated.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier de Valenciennes, Valenciennes, Hauts-de-France, France